CLINICAL TRIAL: NCT03175341
Title: Phase I/II Randomized Study to Evaluate the Role of Intravenous Ascorbic Acid Supplementation to Conventional Neoadjuvant Chemotherapy in Women With Breast Cancer
Brief Title: Intravenous Ascorbic Acid Supplementation in Neoadjuvant Chemotherapy for Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Academic Emergency County Hospital Sibiu (Other)
Collaborators: CHU-UCL Namur (site Mont-Godinne), Belgium (Unknown)
Responsible Party: Principal Investigator, Pop Catalin Florin, MD, Principal Investigator, Academic Emergency County Hospital Sibiu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6222/22.03.2017
Record Dates: First submitted 2017-04-29; First posted 2017-06-05 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; ascorbic acid; vitamin C; vitamin supplementation; quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Ascorbic Acid; Drug Therapy; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized Parallel Assignment
Who Masked: Participant
Masking Description: Single Blind (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C Supplement (Experimental): Ascorbic Acid (AA) with neoadjuvant chemotherapy. Participants received an initial loading dose of 1,5 g Ascorbic Acid (i.v in 100 ml sterile water) on Day 1 followed by 0,75g Ascorbic Acid (i.v in 100 ml sterile water) on Day 2-4 at each chemotherapy cycle and concomitant neoadjuvant chemotherapy regimens administered at the choice of treating physician.
  Ascorbic Acid is administered intravenously before neoadjuvant therapy in D1
  Interventions: Drug: Ascorbic Acid
- Placebo (Active Comparator): Placebos (normal saline (0.9%) with neoadjuvant chemotherapy. 100 ml normal saline 0.9% (placebo) will be administered (i.v) by the same scheme as Ascorbic Acid on Day 1 and respectively Day 2-4 at each chemotherapy cycle.
  Concomitant neoadjuvant chemotherapy regimens administered at the choice of treating physician.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ascorbic Acid — 1,5 g ascorbic acid dissolved in 100 ml sterile water, and 0,75 g ascorbic acid dissolved in 100 ml sterile water.
  Other Names: Vitamin C; Chemotherapy
  Arms: Vitamin C Supplement
Drug: Placebos — 100 ml normal saline 0.9%
  Other Names: Normal Saline; Saline 0.9%
  Arms: Placebo

SUMMARY:
Forty years ago clinical studies conducted by Ewan Cameron and Linus Pauling suggested that intravenous (IV) and oral ascorbic acid (AA) may diminish symptoms and could improve survival in terminal cancer patients. Previous phase I and II clinical trials have found that high dose (1.5g/kg ) iv AA is well tolerated in cancer patients. This is a phase I/II, randomized study of parenteral administration of Ascorbic Acid (AA) as a supplement to the conventional neo-adjuvant chemotherapy in women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score ≤2;
* Diagnosed high-risk breast cancers (tumours ≥ 2cm and/or locally advanced breast tumors) and scheduled to receive neoadjuvant chemotherapy;
* Agree to avoid any additional supplemental ascorbic acid throughout the study;
* Normal glucose-6- phosphate dehydrogenase (G6PD) activity;
* Normal renal function (serum creatinine ≤ 1.2 mg/dl) and normal liver function;
* No evidence of urolithiasis;
* No evidence of chronic hemodialysis, iron overload (serum ferritin 500 ng/ml);
* Not pregnant or lactating women

Exclusion Criteria:

* Important psychosomatic diseases or known gastrointestinal disorders (ulcer, gastritis, colitis, ileitis);
* Current smoking and/or alcohol consumption ≥ 3UI per day;
* Current use of the following drugs:

Aspirin (exceeding 325 mg/day) Acetaminophen (exceeding 2 g/day) Glutathione Vitamin D (important doses)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patients With Adverse Events as a Measure of Safety and Tolerability | during the six months of neoadjuvant chemotherapy
  Assessments are made through analysis of reported incidence of treatment-emergent Adverse Events. Toxicities (AEs) in both groups will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03

SECONDARY OUTCOMES:
Quality of life | At baseline and each 28 days during the six months of neoadjuvant chemotherapy
  The symptom checklist and the symptom related measures as defined by European Organization for Research and Treatment of Cancer (Questionnaire C30 and BR23) will be compared between arms using frequency tables
Therapeutic efficacy | Approximately 6 months
  Therapeutic efficacy assessed by Pathological response. Percentage of Participants Achieving Complete Response (CR) According to the Residual Cancer Burden score.
Objective Response Rate | every 8 weeks, up to 6 months
  Objective Response Rate using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Guidelines
Effect of AA supplementation on serum inflammatory cytokine | At baseline and every 8 weeks during the six months of neoadjuvant chemotherapy
  Assessment of laboratory parameters including interleukin (IL)-6 and vascular endothelial growth factor (VEGF).

CONTACTS AND LOCATIONS:
Overall Officials: Florin Grosu, MD,PhD, Study Director — Academic Emergency County Hospital Sibiu
Locations (1):
- Academic Emergency County Hospital Sibiu, Sibiu, Romania

IPD SHARING:
Plan to Share IPD: No